CLINICAL TRIAL: NCT05588440
Title: Phase 1/2 Multi-Center Study to Evaluate the Safety and Efficacy of ONCT-808 in Adult Subjects With Relapsed or Refractory Aggressive B-Cell Malignancies
Brief Title: A Clinical Study of ONCT-808 in Subjects With Relapsed or Refractory B-Cell Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on the available clinical data and capital requirements for continued development, the Company has decided to terminate this study.
Sponsor: Oncternal Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONCT-808-101
Record Dates: First submitted 2022-09-23; First posted 2022-10-20 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Relapsed/Refractory Aggressive B-Cell Malignancies
Keywords: Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle Cell; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, Non-Hodgkin; ROR1; CAR-T cell therapy; Autologous CAR-T cell therapy; Adoptive cellular therapy; Cellular immunotherapy
MeSH Terms: conditions — Recurrence; Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Dose Escalation (Experimental): Patients will receive a conditioning regimen of cyclophosphamide and fludarabine intravenously (IV) followed by ONCT-808 IV infusion escalated sequentially with a target dose consistent with the dose required by cohort being enrolled to determine Phase 2 dose (RP2d) regimen(s). Participants may receive bridging therapy that is appropriate to the subject's disease and treatment history if clinically indicated to maintain disease stability.
  Interventions: Biological: ONCT-808; Drug: Bridging Therapy
- Phase 2: Dose Expansion (Experimental): Patients with LBCL or MCL will receive ONCT-808 for each RP2D regimen determined in Phase 1.
  Interventions: Biological: ONCT-808; Drug: Bridging Therapy

INTERVENTIONS:
Biological: ONCT-808 — A single infusion of ONCT-808 autologous CAR-T cell infusion will be administered intravenously
  Phase 1: Dose Escalation with bridging therapy as needed
  Phase 2: Patients with LBCL or MCL will be enrolled into two separate dose expansion cohorts.
Drug: Bridging Therapy — Bridging therapy can be oral chemotherapy or IV radiotherapy/chemotherapy per institution's guidelines

SUMMARY:
This is a Phase 1/2 study to investigate the safety and efficacy of the CAR-T therapy, ONCT-808, in patients with relapsed/refractory (R/R) aggressive B cell malignancies.

DETAILED DESCRIPTION:
Study ONCT-808-101 is a Phase 1/2, single-arm, open-label, multi-center study to evaluate the safety and tolerability, pharmacokinetics, and anti-tumor activity of ONCT-808 in subjects with aggressive B cell lymphoma (BCL), including large B-cell lymphoma (LBCL) and mantle cell lymphoma (MCL). The study will be separated into two distinct phases designated as Phase 1 and Phase 2.

After the safety and tolerability of ONCT-808 have been assessed to select the recommended Phase 2 dose (RP2D) in Phase 1, Phase 2 will commence to further validate the dose and evaluate the safety and efficacy of ONCT-808. In Phase 2, subjects with LBCL or MCL will be enrolled into 2 separate dose expansion cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Over 18 years old
* Histologically confirmed aggressive B-cell NHL, including:

  * MCL, with diagnosis confirmed by cyclin D1 overexpression or evidence of t (11;14) translocation
  * LBCL, including:

    * DLBCL NOS
    * Primary mediastinal LBCL
    * High-grade BCL
    * DLBCL arising from follicular lymphoma
    * Follicular lymphoma grade 3B
    * Richter's syndrome
* Availability of archival tissue for immunohistology, or willing to undergo baseline biopsy if not available
* R/R with no available therapy. Subject must have:

  * Received prior systemic therapy that has included an alkylating agent, anthracycline, and an anti-CD20 mAb
  * Received and progressed after autologous hematopoietic stem cell transplant (HSCT) or is ineligible for or has refused to receive HSCT
  * Received prior approved CD19 CAR T-cell therapy or is ineligible for or has refused CD19 CAR-T
* Minimum washout period between previous systemic therapy and leukapheresis includes:

  * Chemotherapy: at least 14 days or 5 half-lives, whichever is shorter
  * Autologous HSCT: at least 3 months
  * CD19 CAR T-cell therapy: at least 6 months
* ≥1 measurable lesion per Lugano criteria (Cheson, 2014)
* Subject has Fluorodeoxyglucose (FDG)-avid disease.
* Subject has an ECOG performance status of 0 or 1.
* Subject has adequate organ function:

  * ALC ≥100/uL
  * ANC ≥1000/uL (≥500/uL if due to lymphoma; growth factors allowed)
  * Hgb ≥8 g/dL (transfusion allowed)
  * Platelets ≥75,000/uL (≥50,000/uL if due to lymphoma; transfusion allowed)
  * CrCL ≥50 ml/min; AST/ALT ≤2.5x ULN, T. bili ≤1.5 mg/dl (except Gilbert's)
  * EF ≥50% by ECHO/MUGA; NCS ECG, NCS pleural effusion; O2 sat >92%
* Subject has an estimated life expectancy of >12 weeks

Key Exclusion Criteria:

* Prior ROR1-targeted therapy
* Current or anticipated systemic immunosuppressive therapy (e.g., prednisone >5 mg) from LD chemo until Day 28 post ONCT-808 dosing
* If receiving anticoagulation therapy, subject is unable to hold therapy for 3 days prior and 28 days following ONCT-808 administration
* Known CNS involvement by malignancy within 6 months
* H/o or current CNS disorder (e.g., seizure, CVA, dementia, cerebellar disease, cerebral edema, posterior reversible encephalopathy syndrome or any autoimmune disease with CNS involvement) within 6 months of study entry
* Clinically significant cardiovascular disease (e.g., MI, UA, CABG, or CHF grade ≥2 NYHA within 12 months of planned ONCT-808 dosing) or serious arrhythmia requiring medication
* Evidence of HIV infection or active HBV, HCV
* Systemic fungal infection requiring medication in the last 12 months
* H/o Covid-19 infection with residual lung infiltrate/fibrosis
* H/o other malignancy except non-melanoma skin cancer or carcinoma in situ not in remission for ≥2 years
* H/o autoimmune disease resulting in end organ injury or require systemic immunosuppression within last 2 years
* H/o allogeneic HSCT or organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wang, Principal Investigator — MD Anderson; Matthew Wei, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: On September 12, 2024, Oncternal Therapeutics, Inc. announced its decision to discontinue the clinical trial evaluating ONCT-808, its ROR1-targeting autologous CAR T program for the treatment of patients with aggressive B-cell lymphoma. The study only enrolled the first few patients into the Phase 1 portion of the study and did not reach a RP2D recommendation. Hence, the Phase 2 portion of the study was not conducted.
Groups:
- ONCT-808 1x10^6 CAR T Cells/kg; ONCT-808 3x10^6 CAR T Cells/kg; ONCT-808 0.3x10^6 CAR T Cells/kg: ONCT-808 consists of autologous CD3/CD28 activated CD4 and CD8 T cells transduced with lentivirus vector expressing a chimeric antigen receptor (CAR) containing a Receptor-tyrosine kinase like Orphan Receptor 1 (ROR1)-directed scFv from zilovertamab (humanized antibody previously known as cirmtuzumab or UC-961) with 4-1BB and CD3 ζ signaling domains
Period: Overall Study
Arm/Group | ONCT-808 1x10^6 CAR T Cells/kg | ONCT-808 3x10^6 CAR T Cells/kg | ONCT-808 0.3x10^6 CAR T Cells/kg
Started | 3 | 2 | 4
Received ONCT-808 One-time Infusion | 3 | 1 | 2
Completed | 0 | 0 | 0
Not Completed | 3 | 2 | 4
Not completed — Sponsor Decision | 2 | 0 | 1
Not completed — Death | 1 | 1 | 1
Not completed — Screen Fail | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ONCT-808 1x10^6 CAR T Cells/kg | ONCT-808 3x10^6 CAR T Cells/kg | ONCT-808 0.3x10^6 CAR T Cells/kg | Total
Number analyzed (Participants) | 3 | 2 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4 | 8
  >=65 years | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 3 | 1 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 2 | 2 | 6
  Hispanic | 1 | 0 | 0 | 1
  Unknown | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Incidence of Dose Limiting Toxicities (DLT)
Description: This is based on subject treated with ONCT-808. ONCT-808 1x10^6 CAR T cells/kg: n=3 ONCT-808 3x10^6 CAR T cells/kg: n=1 ONCT-808 0.3x10^6 CAR T cells/kg: n=2
Time Frame: Up to 28 days after the one-time infusion of ONCT-808
Population: DLT-evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | ONCT-808 1x10^6 CAR T Cells/kg | ONCT-808 3x10^6 CAR T Cells/kg | ONCT-808 0.3x10^6 CAR T Cells/kg
Number analyzed (Participants) | 3 | 1 | 2
Participants | 0 | 1 | 0

2. Secondary Outcome: Best Metabolic Response Rate Post-Baseline
Description: This is based on subject treated with ONCT-808. ONCT-808 1x10^6 CAR T cells/kg: n=3 ONCT-808 3x10^6 CAR T cells/kg: n=1 ONCT-808 0.3x10^6 CAR T cells/kg: n=2
  Response assessments were evaluated using fluorodeoxyglucose (FDG) positron-emission tomography-computed tomography (PET-CT) per the Lugano classification (Cheson, 2014)
Time Frame: up to 1 year after the one-time infusion of ONCT-808
Population: Efficacy evaluable population
Measure: Count of Participants; unit: Participants
Arm/Group | ONCT-808 1x10^6 CAR T Cells/kg | ONCT-808 3x10^6 CAR T Cells/kg | ONCT-808 0.3x10^6 CAR T Cells/kg
Number analyzed (Participants) | 3 | 1 | 2
Participants
  Complete Metabolic Response | 2 | 0 | 0
  Partial Metabolic Response | 1 | 0 | 0
  Not Done (i.e., response assessment was not conducted) | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: AEs collected within 1 year from the date of the one-time infusion of ONCT-808.
Arm/Group | ONCT-808 1x10^6 CAR T Cells/kg | ONCT-808 3x10^6 CAR T Cells/kg | ONCT-808 0.3x10^6 CAR T Cells/kg
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/1 | 1/2
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ONCT-808 1x10^6 CAR T Cells/kg (N=3) | ONCT-808 3x10^6 CAR T Cells/kg (N=1) | ONCT-808 0.3x10^6 CAR T Cells/kg (N=2)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial Spesis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 1 (2) | 1 (1) | 0 (0)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encenphalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ICANS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Systolic Dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ONCT-808 1x10^6 CAR T Cells/kg (N=3) | ONCT-808 3x10^6 CAR T Cells/kg (N=1) | ONCT-808 0.3x10^6 CAR T Cells/kg (N=2)
Cytokine Release Syndrome (Immune system disorders) | 2 (5) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT05588440/Prot_SAP_002.pdf